CLINICAL TRIAL: NCT05276479
Title: Association Between Dietary Plant Hormone Intake and Mental Health
Brief Title: Dietary Plant Hormone and Mental Health
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: ABA2022
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Dietary Behavior; Stress; Sleep; Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mental Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects: Healthy subjects aged 18-30 years
  Interventions: Other: Anonymous online survey on dietary habits and mental health

INTERVENTIONS:
Other: Anonymous online survey on dietary habits and mental health — Assessment of regular feeding behavior and mental health

SUMMARY:
The aim of this cross-sectional online study is to investigate the association between regular feeding behavior and stress, sleep as well as anxiety and depressive symptoms in healthy subjects.

DETAILED DESCRIPTION:
The gut-microbiota-brain (GMB) axis has a multidirectional communication between the intestine, the microbiota, and the central nervous system (CNS). Over the past decade, there has been extensive research showing that the GMB axis has a profound influence not only on neurological disorders but also on neural development, activation of the neuroendocrine axis and neurotransmission, as well as modulation of complex human behaviors. Thus, the GBM-axis is involved in the regulation of stress, emotions, behaviour, and higher cognitive functions. As the GMB plays an essential role in human psychological functioning and mental health, the dietary manipulation of the microbiome may have direct effects on mental well-being, sleep, anxiety and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 30

Exclusion Criteria:

* None

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Mental well-being and quality of life | At baseline
  Subjective life-quality will be measured with the short version of the World Health Organization Quality of Life questionnaire (WHOQOL-BREF,). The WHOQOL-BREF is a self-administered questionnaire comprising 26 questions on the individual's perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely". For the present study only the three subscales (physical and psychological health, and social relationships) will be assessed.
General Psychopathology | At baseline
  Brief Symptom Checklist (BSCL former BSI), including various subscales such as depression, anxiety
Sleep | At baseline
  Sleep quality is assessed with the Pittsburgh Sleep Quality Index (PSQI). Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.

SECONDARY OUTCOMES:
Stress and Coping | At baseline
  Stress will be assessed with the Stress and Coping Inventory (SCI).The SCI is used to determine the current stress load and stress symptoms and to illustrate how to deal with stress using five coping strategies. It comprises 10 scales with 54 items: (A) Current stress load (1) Stress due to uncertainty, (2) Stress due to overload, (3) Stress due to loss and actual negative events, (4) Total stress: Total stress due to insecurity, threat, overload or loss in important areas of life, (5) Physical and psychological stress symptoms; (B) Stress coping (Coping) (1) Positive thinking, (2) Active stress coping, (3) Social support, (4) Keeping faith, (5) Increased alcohol and cigarette consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Leila M Soravia, Prof. Dr., Principal Investigator — University Hospital of Psychiatry, University of Bern
Locations (1):
- University Hospital of Psychiatry, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No